CLINICAL TRIAL: NCT01258751
Title: A Phase 1, Open-Label Study To Evaluate 5-Ht6 Receptor Occupancy As Measured By Positron Emission Tomography (PET) With Ligand [11c]PF-04171252 Following Single Oral Dose Administration Of PF-05212377 (Sam-760) In Healthy Subjects
Brief Title: This Study Will Evaluate The Relationship Between Plasma Drug Levels And Receptor Binding In Brain Using PET (Positron Emission Tomography) In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Yale University (Other)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B2081007; B2081007
Record Dates: First submitted 2010-12-09; First posted 2010-12-13 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-07

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — SAM-760

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-05212377 (Experimental)
  Interventions: Drug: PF-05212377

INTERVENTIONS:
Drug: PF-05212377 — Single dose of up to 70 mg PF-05212377, delivered as .25 mg, 5 mg and/or 15 mg on study day 1
  Other Names: SAM-760

SUMMARY:
The purpose of this study is to evaluate the relationship between plasma drug levels and receptor binding in brain using PET; and to evaluate safety and tolerability after a single administration of PF-05212377 in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of nonchildbearing potential between the ages of 18 and 55 years, inclusive

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening
* Fulfillment of any of the MRI contraindications on the standard radiography screening questionnaire

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To assess the central 5-HT6 receptor occupancy (RO) in the striatum in relation to systemic exposure of PF-05212377 after single oral administration in healthy adult subjects. | up to 8 days

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | continuous, up to 8 days
Maximum concentration (Cmax) for PF-05212377 in plasma | up to 8 days
Time at Cmax (Tmax) for PF-05212377 in plasma | up to 8 days
Area under the concentration-time profile from time zero to the time of the last quantifiable concentration (AUClast) for PF-05212377 in plasma | up to 8 days
Average concentration during the first post-dose PET scan (Cavg (scan 1)) for PF-05212377 in plasma | approximately 4-6 hrs post-dose
Average concentration during the second post-dose PET scan (Cavg (scan 2)) for PF-05212377 in plasma | approximately 28-30 hrs post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Sawant-Basak A, Chen L, Lockwood P, Boyden T, Doran AC, Mancuso J, Zasadny K, McCarthy T, Morris ED, Carson RE, Esterlis I, Huang Y, Nabulsi N, Planeta B, Fullerton T. Investigating CNS distribution of PF-05212377, a P-glycoprotein substrate, by translation of 5-HT6 receptor occupancy from non-human primates to humans. Biopharm Drug Dispos. 2023 Feb;44(1):48-59. doi: 10.1002/bdd.2351. Epub 2023 Mar 13. PMID 36825693
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2081007&StudyName=This%20Study%20Will%20Evaluate%20The%20Relationship%20Between%20Plasma%20Drug%20Levels%20And%20Receptor%20Binding%20In%20Brain%20Using%20PET%20%28Positron%20Emission%20Tomogr